CLINICAL TRIAL: NCT06336408
Title: Explore the Effects of SLEEP Deprivation on Short-term Outcomes in ICU pAtients basEd on polysomnogRaphy：a Single-center Prospective Cohort Study
Brief Title: The SLEEP-CARE Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2023-370R
Record Dates: First submitted 2024-03-13; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-01

CONDITIONS: Sleep Disturbance
Keywords: Polysomnography; intensive care unit
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sleep disorder is common in ICU patients, such as reduced sleep time, fragmentation, and abnormal sleep rhythm. In 2023, American Thoracic Society released a research statement on sleep and circadian disruption(SCD) in ICU, which considered SCD is an important potential target for improving critical illness outcomes. Although polysomnography(PSG) is the gold standard of sleep measurement, subjective sleep evaluation tools are still used in most clinical studies related to sleep in ICU. This makes the sleep quality of ICU patients overestimated and difficult to reflect their true sleep conditions. And the answers to how and which outcomes different levels of sleep deprivation affect patient outcomes are still unclear and need to be further explored.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥ 18-years old)
* anticipated SICU stay for 24 hours or more

Exclusion Criteria:

* pregnancy
* Have a clear history of medication for sleep disorders
* History of mental or psychological illness
* Treated with CRRT or ECMO during monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Compound outcome index | Discharge from ICU or 2 weeks
  Patients with cognitive, respiratory, digestive, cardiovascular, or immune-related adverse outcomes. Cognitive-related adverse outcomes were defined as delirium in the ICU(using Confusion Assessment Method Intensive Care Unit to screen delirium as negative or positive). Respiratory-related adverse outcomes was defined as a decrease in blood gas oxygenation index below 300mmHg in ICU. Gastrointestinal related adverse prognosis was defined as bleeding from stress ulcer in ICU. Cardiovascular-related adverse outcomes were defined as newly diagnosed heart failure, arrhythmia, and myocardial infarction in ICU. Immune-related poor prognosis defined SOFA (Sequential Organ Failure Assessment) scores increased by more than 2 points compared to the time of entry.

SECONDARY OUTCOMES:
LOS | Through study completion, an average of 10 days
  length of ICU stay

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China